CLINICAL TRIAL: NCT01657071
Title: A Randomized, Open-label, Single Dose, 2-treatment, 2-period, 2-way Crossover Study to Assess the Pharmacokinetic Characteristics of YH14659, a Fixed Dose Combination Compared With Coadministration of Separate Constituents Under Fasted Conditions in Healthy Male Subjects
Brief Title: Comparative Pharmacokinetics of YH14659 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH14659-102
Record Dates: First submitted 2012-03-21; First posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: YH14659
- Group B (Active Comparator)
  Interventions: Drug: clopidogrel & aspirin

INTERVENTIONS:
Drug: YH14659 — YH14659 capsule by oral
  Arms: Group A
Drug: clopidogrel & aspirin — clopidogrel tablet(75mg) + aspirin capsules(100mg) by oral
  Arms: Group B

SUMMARY:
The objective of this study is to compare pharmacokinetics after single oral administration of 2 capsules of YH14659, a fixed-dose combination of clopidogrel and aspirin developed by Yuhan Corporation versus co-administration of Plavix (clopidogrel) and Astrix (aspirin) in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers of aged between 20 years to 55 years
* Weight: over 50kg, within ±20% of ideal body weight
* Have no history of neither congenital nor chronic disease
* Have no history of abnormal symptoms or opinions as a result of physical examination (medical checkup)
* Eligible subjects with acceptable medical history, physical examination, laboratory tests, ECG during screening period
* Subject who has signed on the written consent

Exclusion Criteria:

* Have a known allergy or hypersensitivity to anti-platelet agents
* Person with hypotension (SBP ≤ 100mmHg or DBP ≤ 50mmHg) or hypertension (SBP ≥ 150mmHg or DBP ≥ 95mmHg), person whose pulse rate is below 45 or over 100 a minute
* Have the following abnormal findings on diagnosis;

  * have AST or ALT > 1.25 times of normal upper limit
  * have total bilirubin > 1.5 times of normal upper limit
  * have higher PT, aPPT, BT than normal range
  * have PLT below 180,000 or above 350,000
* Patients with hemorrhage or predisposition to hemorrhage
* Have disease or history of stomach or intestinal surgery or resection that would potentially alter absorption of orally administered drugs
* Have participated in other clinical studies within 3 months prior to the first administration
* Have used any prescription medications including anti-coagulants, anti-platelet agents, thrombolytic drugs and Prostaglandin E1 agents within 2 weeks prior to the first administration or any over-the-counter, non-prescription preparations within 1 week prior to the first administration
* Patients with aspirin induced asthma(AIA) or history of AIA
* Subject who is judged to be ineligible by principal investigator or sub-investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Cmax and AUCt of clopidogrel | 24hrs
Cmax and AUCt of Acetylsalicylic acid | 24hrs

SECONDARY OUTCOMES:
Tmax, T1/2, λz and AUC∞ of Clopidogrel and Acetylsalicylic acid - AUCt, Cmax, Tmax, T1/2, λz and AUC∞ of salicylic acid | 24hrs
AUCt, Cmax, Tmax, T1/2, λz and AUC∞ of salicylic acid | 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: Jang-Hee Hong, M.D., Ph.D., Principal Investigator — Chung-Nam National University Hospital
Locations (1):
- Yuhan Corporation, Seoul, South Korea